CLINICAL TRIAL: NCT01714700
Title: Interactive Effects of an Isocaloric High-protein Diet and Resistance Exercise on Body Composition, Ghrelin, and Metabolic and Hormonal Parameters in Untrained Overweight Young Men
Brief Title: Interactive Effects of an Isocaloric High-protein Diet and Resistance Exercise in Untrained Overweight Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GHRELIN0912
Record Dates: First submitted 2012-10-18; First posted 2012-10-26 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Overweight; Obesity
Keywords: protein; resistance exercise ghrelin; overweight
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet, High-Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High protein diet, Resistance exercise (Active Comparator): High protein diet, Resistance exercise total calories 2400 Kcal/day, 55% carbohydrate, 30% protein, and 15% fat
  Interventions: Behavioral: High protein diet, Resistance exercise; Behavioral: Standard diet, Resistance exercise
- Standard diet, Resistance exercise (Placebo Comparator): total calories 2400 Kcal/day, 60% carbohydrate, 15% protein, and 25% fat; ST group
  Interventions: Behavioral: High protein diet, Resistance exercise; Behavioral: Standard diet, Resistance exercise

INTERVENTIONS:
Behavioral: High protein diet, Resistance exercise — The progressive supervised resistance exercise training program was performed by all participants under supervision. They participated in an onsite supervised protocol for 12 weeks (six days per week); weeks 1-4 (Monday - pectorialis major, Tuesday - latissimus dorsi, Wednesday - femoral, Thursday - deltoid, Friday - biceps brachii, Saturday - triceps brachii muscle), weeks 5-8 (Monday and Friday- pectorialis major and triceps brachii, Tuesday and Saturday - latissimus dorsi and biceps brachii, Wednesday and Monday - femoral, Thursday and Tuesday - deltoid muscle), weeks 9-12 (Monday and Thursday - pectorialis major and latissimus dorsi, Tuesday and Friday - femoral and deltoid, Wednesday and Saturday - triceps brachii and biceps brachii muscle).
Behavioral: Standard diet, Resistance exercise — The progressive supervised resistance exercise training program was performed by all participants under supervision. They participated in an onsite supervised protocol for 12 weeks (six days per week); weeks 1-4 (Monday - pectorialis major, Tuesday - latissimus dorsi, Wednesday - femoral, Thursday - deltoid, Friday - biceps brachii, Saturday - triceps brachii muscle), weeks 5-8 (Monday and Friday- pectorialis major and triceps brachii, Tuesday and Saturday - latissimus dorsi and biceps brachii, Wednesday and Monday - femoral, Thursday and Tuesday - deltoid muscle), weeks 9-12 (Monday and Thursday - pectorialis major and latissimus dorsi, Tuesday and Friday - femoral and deltoid, Wednesday and Saturday - triceps brachii and biceps brachii muscle)

SUMMARY:
Background: The interactive effects of resistance training and dietary protein on hormonal responses in overweight or obese adults are not clear and remain controversial. Investigators tested the effect of an isocaloric high-protein diet on body composition, ghrelin, and metabolic and hormonal parameters during a 12-week resistance training program in untrained overweight healthy young men.

Methodology: Investigators randomized 18 healthy young males to a standard diet (ST group) or an isocaloric high protein diet (HP group). Subjects in both groups participated in a 12 week-resistance exercise program. Investigators measured body composition, lipid profile, homeostatic model assessment of insulin resistance (HOMA-IR) indices, total ghrelin, and exercise related hormones at baseline and 12 weeks.

DETAILED DESCRIPTION:
Background: The interactive effects of resistance training and dietary protein on hormonal responses in overweight or obese adults are not clear and remain controversial. Investigators tested the effect of an isocaloric high-protein diet on body composition, ghrelin, and metabolic and hormonal parameters during a 12-week resistance training program in untrained overweight healthy young men.

Methodology: Investigators randomized 18 healthy young males to a standard diet (ST group) or an isocaloric high protein diet (HP group). They have not participated in any weight-management program during the previous 6 months. An open-label design will be used. At enrolment, participants will randomly assign to one of two groups: a control group with a standard diet (total calories 2,400 kcal/day, 60% carbohydrate, 15% protein and 25% fat; ST group) and an interventional group with an isocaloric high protein diet (total calories 2,400 kcal/day, 55% carbohydrate, 30% protein and 15% fat; HP group). Participants in both groups take part in a scheduled resistance exercise training program. Participants does not take part in any other resistance training program or competitive sport over the study duration. At the start of the study, participants will be instructed to maintain their assigned diet throughout the study period. This will be assessed using a food frequency questionnaire (FFQ) with a 24-h recall after 12 weeks. Participants are presented with two-dimensional food pictures of the actual size of portions on a computer by a single trained dietitian to minimize interviewer bias. Medium are defined as the portion sizes shown, small are approximately half the medium portion size, and large are one-and-a-half times the medium portion size.

Exercise Protocol All participants will be under supervision during participation in the progressive supervised resistance exercise-training program. They participate in an onsite supervised protocol for 12 weeks (6 days per week). Exercise duration will be increased gradually, from 50 min at week 1 to 80 min at week 12, including warm-up for 20 min and cool-down periods for 10 min by carrying out gentle stretching exercises of the upper and lower limbs. A one repetition maximum (1-RM) is the maximum weight that can be lifted for one complete repetition of the movement. For each participant, the RM will be calculated for a particular muscle group. Each movement will be carried out at 60-80% of his 1-RM. Resistance will be increased slowly by three steps; step 1 (60-70% of his 1-RM for week 1-4), step 2 (65-75% of his 1-RM for week 5-8) and step 3 (70-80% of his 1-RM for week 9-12).

Baseline and Follow-up Measurements Height and bodyweight are measured using a digital scale with the examinee wearing a light gown, but no shoes. Body mass index (BMI) are calculated as weight (kg) divided by height squared (m2). The percentage body fat and total fat mass are measured by bioelectric impedance analysis (Inbody 3.0; Biospace Co., Ltd., Seoul, Korea), a sensitive test for quantification of changes in lean and fat mass in vivo and for assessment of regional fat distribution. A mercury sphygmomanometer are used for measurement of blood pressure (BP) of each participant, in the sitting position, after a 10-min resting period. Two readings each for the systolic and diastolic Bps are recorded at 3-min intervals, and the average of each measurement are included in our analysis.

Blood samples are obtained preprandially at 0.800 hours from each participant's antecubital vein after a 12-h fast, and are used for determination of plasma glucose, insulin, lipid profile, total ghrelin, GH, insulin-like growth factor-1 (IGF-1), testosterone and cortisol. Blood samples are obtained at baseline (prerandomization) and 12 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

- Eighteen healthy young males overweight

Exclusion Criteria:

- participated in any weight-management program during the previous six months

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-08; Primary Completion 2007-03 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
body composition | 12-week
  BMI, and body fat percent

SECONDARY OUTCOMES:
ghrelin | 12-week
  ghrelin
Insulin resistance | 12-week
  HOMA-IR
lipid parameter | 12-week
  lipid
growth hormone | 12-week
  GH, IGF-1
hormone | 12-week
  testosterone
cortisol | 12-week
  cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Pusan, Ami-dong, South Korea

REFERENCES:
- [Derived] Kim HH, Kim YJ, Lee SY, Jeong DW, Lee JG, Yi YH, Cho YH, Choi EJ, Kim HJ. Interactive effects of an isocaloric high-protein diet and resistance exercise on body composition, ghrelin, and metabolic and hormonal parameters in untrained young men: A randomized clinical trial. J Diabetes Investig. 2014 Mar 23;5(2):242-7. doi: 10.1111/jdi.12148. Epub 2013 Oct 10. PMID 24843767